CLINICAL TRIAL: NCT03694977
Title: Biomarker Study of PDR001 in Combination With MCS110 in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yung-Jue Bang, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1710-062-893
Record Dates: First submitted 2018-09-19; First posted 2018-10-03 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: MCS110/PDR001 combination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCS110/PDR001 combination (Experimental)
  Interventions: Drug: MCS110/PDR001 combination

INTERVENTIONS:
Drug: MCS110/PDR001 combination — MCS110 7.5mg/kg iv since 1st cycle PDR001 300 mg iv since 2nd cycle Q 3weeks

SUMMARY:
<Background>

1. Current status of treatment options in advanced gastric cancer.

   * The cytotoxic chemotherapy, usually fluoropyrimidine + platinum combination regimen is current standard of care. In case of HER2(+) gastric cancer, the addition of trastuzumab on top of cytotoxic chemotherapy is standard of care.
   * In second-line setting, the cytotoxic chemotherapy in combination with Ramucirumab improved the patients' survival compared with cytotoxic chemotherapy alone.
   * There are few treatment options for gastric cancer patients who have been treated with more than two lines of palliative chemotherapy. Patients with good performance status even after failure to 2 kinds of palliative chemotherapy still need the active anticancer treatment options. Therefore, this is the high unmet medical need.
2. Current status of immunotherapy development in gastric cancer
3. The importance of tumor microenvironment
4. The role of polarized macrophage in TME
5. The role of polarized macrophage in gastric cancer
6. Potential of combination of PD1 inhibitor and CSF-1 inhibitor

Based on these rationales, we hypothesized that the combination of PD1 inhibitor and CSF1R inhibitor might be synergistic in gastric cancer. However, the exact in vivo immune modulation by each inhibitor has not been revealed so far. Therefore, we will conduct this "biomarker study of PDR001 in combination with MCS110 in gastric cancer" to see the biologic dynamic modulation with MCS110 and combination (MCS110/PDR001) and to see preliminary efficacy signal with this combination.

<Trial objectives> Primary objective: To see biomarker changes (PDL1, TAM, TIL) by MCS110 monotherapy and MCS110/PDR001 combination (To see the biomarker changes by MCS110 monotherapy at first, then, by MCS110/PDR001 combination in gastric cancer) Secondary objective: To see preliminary efficacy (ORR, irRR, PFS, DOR, DCR, OS) and safety.

DETAILED DESCRIPTION:
<Background>

1. Current status of treatment options in advanced gastric cancer.
2. Current status of immunotherapy development in gastric cancer

   * Harnessing immune system to fight against cancer cells is one of highlighting strategy in new drug development in almost all kinds of solid tumor including gastric cancer.
   * In PD L1expressing gastric cancer, the anti-PD1 antibody monotherapy (pembrolizumab) shows the antitumor efficacy. (Bang YJ et al. 2015)
   * Anti-PDL1 antibody (Avelumab) used in the first-line maintenance setting or 2nd-line setting of biomarker-unselected gastric cancer also shows promising antitumor efficacy (Chung HC et al. ECCO/ESMO 2015, Oh DY et al. ASCO GI 2016)
   * There are many clinical trials using immune-oncology (IO) agents are ongoing in 1st-line setting, 2nd-line setting, 3rd-line setting and refractory setting. Several strategies are being used, that is, IO monotherapy in biomarker-selected population, IO+IO combination, IO+cytotoxic chemotherapy , and IO+other targeted agents to improve the efficacy of harnessing immune system.
   * Still, we don't know the exact biomarker for these IO agents in gastric cancer. Not all patients get the benefit with these agents.
3. The importance of tumor microenvironment

   * From the immunotherapy point of view, the tumor microenvironment (TME) should be considered for the successful immunotherapy.
   * In TME, many components working for antitumor immunity and intratumoral immunosuppression exist. (Pitt JM et al. 2016)
   * The most crucial and direct control of tumor cells is performed by CD4+ T helper cell and CD8+ cytotoxic T lymphocyte (CTL). Th1 response, characterized by T cell production of IFN-ɣ, TNF-α, IL-2 are considered to be the essential subset for tumor rejection. However, Th1 response also contributes to tumor escape via IFN-ɣ-mediated expression of the inhibitory checkpoint molecules PDL1 or via the selection of resistant clones through tumor immunoediting.
   * Long-term exposure to tumor antigen induces Th1 cells and other T cells that lack the typical poly-functional phenotype and that express inhibitory receptors such as PDL1. LAG-3, and TIM-3.
   * Other subsets of CD4+T cells inhibit antitumor immune responses. CD4+Tregs is the example. Tregs inhibit the antitumor activity of CTLs and NK cells either directly, or indirectly via APCs. In addition to Tregs, Th2 cells can also block Tcell-induced tumor rejection.
   * TME can also directly impair intratumoral T cell proliferation, acting as another mechanism for tumor evasion of immune surveillance. IDO production within the TME is the example. IDO produced by myeloid cells and cancer cells catabolizes tryptophan to generate kynurenine, which together promotes the conversion of naïve T cells to Tregs,inhibition of Treg reprogramming to potentially anti-tumoral Th cells, and increases MDSC functions through upregulation of IL-6 expression.
4. The role of polarized macrophage in TME

   * Macrophages are one of the major components of the TME, are recruited by chemokines such as M-CSF and chemokine C-C motif ligand 2, and are produced mainly be tumor cells (Wiktor-Jedrzejczak W, et al. 1996)
   * Macrophages are dynamic cells that can express different functional programs in response to microenvironmental signals (Mantovani A, et al. 2004)
   * Bacterial stimuli, IFN-ɣ and GM-CSF promote a proinflammatory M1-polarized phenotype, whereas M-CSF, IL-4, and IL-13 favor the generation of folate receptor b positive, IL-10 producing, immunosuppressive, M2-polarized macrophages. (Murray PJ, et al. 2011). M1 macrophages also amplify TH1 responses, providing a positive feedback loop in the antitumor response.
   * Macrophages that infiltrate tumor tissues, also termed tumor-associated macrophages (TAMs), can be driven by tumor-derived and T-cell derived cytokines to acquire such a polarized phenotype, and have a key role in subversion of adaptive immunity and in inflammatory circuits that promote tumor growth and progression. (Mantovani A, et al. 2002)
   * Fully polarized M1 and M2 macrophages are the extremes of a continuum of functional states; in contrast to this binary M1/M2 definition, there are several other distinct populations that share features of both types.( Ojalvo LS, et al. 2009)
   * The M2-polarized macrophages promote tumor progression and metastasis by activating circuits that regulate tumor growth, adaptive immunity, stroma formation, and angiogenesis, and can be used as prognostic indicators. ( Balkwill F, et al. 2001)
5. The role of polarized macrophage in gastric cancer

   * In gastric cancer, infiltration of polarized TAMs is an independent prognostic factor. (Zhang, et al. 2015)
   * The number of peritoneal macrophages with the M2 phenotype (CD68+CD163+ or CD68+CD204+) was significantly higher in gastric cancer patients with peritoneal dissemination than in those without peritoneal dissemination. (Yamaguchi et al. 2015)
   * Higher expression of M2-related messenger RNA (IL-10, VEGF-A, VEGF-C, MMP-1, amphiregulin), lower expression of M1-related messenger RNA (TNF-am CD80, CD86, IL-12p40) were confirmed in the TAM of gastric cancer.
   * Interestingly, macrophage co-culture with gastric cancer cells converted M1 phenotype into M2 phenotype. Moreover, the coexistence of MKN45 cells with M2 macrophages resulted in cancer cell proliferation and an acceleration of tumor growth in the xenograft model.
   * In our hospital, we investigated the prognostic significance of TAM in MSI-high gastric cancers using IHC. (Kim et al. 2015) CD68 and CD163 were used as markers for total infiltrating macrophages and M2-polarized macrophages, respectively. The density of CD68+ or CD163+ TAMs in four different areas (epithelial and stromal compartments of both the tumor center and invasive front) were analyzed in 143 cases of MSI-high advanced gastric cancers.

   In multivariate survival analysis, CD163+ TAMs in four combined areas, stromal and epithelial compartments of both tumor center and invasive front were independent prognostic indicator in MSI-high gastric cancers.
   * Polarized CD163+ TAM was also reported to be associated with increased angiogenesis and CXCL12 expression in gastric cancer (Park et al. 2015)
   * We investigated the role of cytokine and angiogenic factors in the gastric cancer (Ock et al. 2015, Ock et al. 2016). High serum level of M-CSF is associated with poor survival outcome in gastric cancer patients who received standard 1st-line chemotherapy.
6. Potential of combination of PD1 inhibitor and CSF-1 inhibitor

   * Blockade of colony-stimulating factor-1 (CSF-1) limits macrophage infiltration and improves response of mammary carcinomas to chemotherapy. ( Ruffell B et al. Cancer Cell 2014)
   * In BRAF mutant melanoma model, CSF1R inhibitor (PLX3397) reduced the recruitment of CD11bC Gr1lo and CD11bC Gr1int M2-like macrophages, but this was accompanied by an accumulation of CD11bC Gr1hi cells. PDL1 expression on remaining myeloid cells potentially dampened the antitumor efficacy of BRAF inhibitor (PLX3397) and PLX4720 in combination, since PD1/PDL1 axis blockade improved outcome. (Ngiow SF et al. 2015)
   * In pancreatic cancer model, inhibiting signaling by the myeloid growth factor receptor CSF1R can functionally reprogram macrophage responses that enhance antigen presentation and productive antitumor T-cell responses. (Zhu Y et al. 2014) However, CSF1R blockade also upregulated T-cell checkpoint molecules, including PDL1 and CTLA4, thereby restraining beneficial therapeutic effects.
   * In these cases, combination of CSF1R blockade and PD1 or CTLA4 inhibitor potently decreased tumor progression.

<Trial design and plan> Each dosing interval will be 3 weeks.

1. Before 1st dosing of MCS110, 1st fresh tumor biopsy will be done.
2. After 1st dosing of MCS110 monotherapy, 2nd fresh tumor biopsy will be done
3. Then, combination of MCS110 with PDR001 will be initiated.
4. After 1st dosing of MCS110/PDR001 combination, 3rd fresh tumor biopsy will be done.
5. After that, the MCS110/PDR001 combination will be delivered to the patients until disease progression, intolerable toxicity, or patient's consent withdrawal.
6. At the time of disease progression, fresh tumor tissue will be obtained if possible (optional).
7. In each tumor biopsy time point, blood sampling will be accompanied.
8. Tumor response evaluation will be done every 2 cycles of MCS110/PDR001 combination treatment.

Translational research that will be performed. The description of biomarker changes will be the main purpose of this biomarker study. Therefore, the translational research is the main interest of this study.

The candidate biomarkers are as below, which was adopted from the MCS110Z2102 clinical trial. However, the exact analysis items will be chosen based on the tumor tissue amount and developing science during study period. The main focus will be on PDL1, TAM, TIL.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female patient, age ≥ 20 years
3. Pathologically confirmed unresectable or recurrent gastric cancer
4. Patients who have previously treated with at least 2 kinds of palliative chemotherapy
5. Patients must have measurable disease by RECIST 1.1
6. Patients must have easily assessable tumor sites for fresh biopsy
7. ECOG performance status of 0-1
8. Adequate bone marrow, organ function and laboratory parameters:

   * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L,
   * Hemoglobin (Hgb) ≥ 8 g/dL without transfusions,
   * Platelets (PLT) ≥ 75 x 109/L without transfusions,
   * AST and ALT ≤ 3 × upper limit of normal (ULN),
   * Total bilirubin ≤ 1.5 × ULN, (Patients with biliary obstruction can join if bilirubin corrects to required limit after adequate biliary drainage)
   * Creatinine ≤ 1.5 mg/dL
9. Adequate cardiac function:

   • QTc interval ≤ 480 ms
10. Negative serum β-HCG test (female patient of childbearing potential only) performed locally within 72 hours prior to first dose.

Exclusion Criteria:

1. Presence of symptomatic CNS metastasis 2 History of severe hypersensitivity reactions to other monoclonal antibodies 3. Impaired cardiac function or clinically significant cardiac disease 4. Active autoimmune disease or a documented history of autoimmune disease within 3 years before screening 5. Active infection, including active tuberculosis requiring systemic antibiotic therapy 6. Known HIV infection 7. Active HBV or HCV infection. HBV carrier without detectable HBV DNA is not excluded 8. Other malignant disease. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment: completely resected basal cell and squamous cell skin cancers: any malignancy considered to be indolent and that has never required therapy, and completely resected carcinoma in situ of any type 9. Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.

10. History of previous immune-related abnormal reaction or current interstitial lung disease, noninfective interstitial lung disease or drug-induced interstitial pneumonitis 11. Patients who failed immune check point inhibitors which includes PD-1, PDL-1, CTLA4 antagonist and investigational drugs.

12. Patients requiring chronic treatment with systemic steroid therapy or any immunosuppressive therapy, other than replacement-dose steroids in the setting of adrenal insufficiency.

13. Use of any live vaccines against infectious disease within 4 weeks of initiation of study treatment.

14. Major surgery within 2 weeks of the first dose of study treatment 15. Radiotherapy within 2 weeks of the first dose of study treatment, except for palliative radiotherapy to a limited field.

16. Systemic chemotherapy within 3 weeks of the first dose of study treatment. In case of mitomycin Cor nitrosoureas, 4 weeks rest should be needed.

17. Presence of ≥ CTCAE Gr2 hematologic toxicity or ≥ CTCAE Gr3 non-hematologic toxicity(except for alopecia) caused by previous chemotherapy 18. Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF, M-CSF) ≤ 2 weeks prior start or study drug. An erythroid stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment.

19. Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 150 days after the last dose of PDR001 or 90 days after the last dose of MCS110 for patients who stopped PDR001 and continued MCS110 alone for more than 60 days.

21. Sexually active males unless they use a condom during intercourse while taking treatment and for150 days after the last dose of PDR001 or 90 days after the last dose of MCS110 for patients who stopped PDR001 and continued MCS110 alone for more than 60 and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of potential biomarkers of MCS110 in combination with PDR001 | 3weeks
  The current study explores potential biomarkers of MCS110 in combination with PDR001 that predict tumor response in the tumor tissue and blood of patients with gastric cancer.

SECONDARY OUTCOMES:
Objective response rate | 6weeks
  According to RECIST v1.1 criteria
Immune-related response rate | 6weeks
  According to RECIST v1.1 criteria
Progression-free survival | 6weeks
  Time from randomization until disease progression or death
Duration of response | 6weeks
  Time from documentation of tumor response to disease progression
Disease control rate | 6weeks
  The percentage of patients who have achieved complete response, partial response and stable disease
Overall survival | 3months
  Time from randomization until death from any cause
Safety as measured by number and grade of toxicity events | 3weeks
  According to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No